CLINICAL TRIAL: NCT06146699
Title: Status of Diabetic Retinopathy and Its Presentation Patterns in Diabetics at Assiut University Hospital
Brief Title: Prevalence of Diabetic Retinopathy in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelhafez Mohamed, Principal Investigator, Assiut University
Other Study IDs: Diabetic Retinopathy
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Tomography, Optical Coherence; Fluorescein Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — Optical Coherence Tomography (OCT) is a non-invasive diagnostic technique that renders an in vivo cross-sectional view of the retina.
Device: Fundus fluorescein angiography (FFA) — Fundus fluorescein angiography (FFA) is an invasive diagnostic procedure. It helps to assess the anatomy, physiology, and pathology of retinal and choroidal circulation. It aids in the diagnosis of various ocular pathologies.

SUMMARY:
To determine the stage of Diabetic Retinopathy (DR) and the presenting symptoms at the time of ophthalmological examination of diabetic individuals .

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the main cause of decreased vision and blindness in patients with diabetes throughout the world . In Egypt, the estimated prevalence of diabetes mellitus (DM) is expected to rise from 5-10% in the 1990s to>13% of the population over 20 years old by 2025 .

The estimation of the prevalence of diabetic retinopathy (DR) is challenging due to the great variation in the study populations, methodologies, and grading schemes .

Globally, the prevalence of DR and diabetic macular edema (DMO) is expected to rise from the estimates for the period 2015-2019 (27%) due to the expected increase in the life expectancy of people living with DM .

Diabetic retinopathy is now the 5th leading cause of blindness worldwide and is the main cause of blindness in working population .

Blindness due to diabetic retinopathy is more common in type 1 diabetics (4%) than in type 2 (1.6%) .

The exact mechanism of how prolonged hyperglycaemia causes retinopathy is still unclear, however studies have shown that prolonged hyperglycaemia alters retinal perfusion thereby disturbing the normal physiological and homeostatic state of the retina, in turn causing retinopathy .

Fortunately, much of the visual loss from DR is preventable, and the rates of vision loss from diabetes and DR have steadily declined over the past few decades. Such improvements in visual outcomes for DR are multifactorial, and are due in large part to a combination of better systemic risk factor control, coupled with advances in ocular disease assessment, screening, imaging and treatment in recent years .

ELIGIBILITY:
Inclusion Criteria:

* All known diabetic patients ( type 2 ) or patients who were later on diagnosed with type 2 diabetes mellitus as per American Diabetes Association (ADA) criteria who presented for the first time to Assuit university hospital opthalomolgy outpatient clinics during study duration (one year) will be included in the study . Diabetic retinopathy will be classified according to Early Treatment Diabetic Retinopathy Study (ETDRS) classification as mild, moderate, severe and very severe non proliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR). Patients with vitreous hemorrhage, rubeosis iridis, neovascular glaucoma or tractional retinal detachment will be classified as having advanced diabetic eye disease (ADED).

Exclusion Criteria:

* Type 1 Diabetic patients or patients with diabetes below 25 years old will be excluded from the study .

Ages: 25 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All known diabetic patients ( type 2 ) or patients who were later on diagnosed with type 2 diabetes mellitus as per American Diabetes Association (ADA) criteria
Sampling Method: Non-Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of diabetic retinopathy | Baseline
  To determine the stage of Diabetic Retinopathy (DR) and the presenting symptoms at the time of ophthalmological examination of diabetic individuals .

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf K. Al-Hussaini, prof, Study Chair — Assiut University; Ahmed M. Fahmy Fathalla, prof, Study Director — Assiut University; Islam M. Mohamed Gouda, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thapa SS, Thapa R, Paudyal I, Khanal S, Aujla J, Paudyal G, Rens Gv. Prevalence and pattern of vitreo-retinal diseases in Nepal: the Bhaktapur glaucoma study. BMC Ophthalmol. 2013 Mar 28;13:9. doi: 10.1186/1471-2415-13-9. PMID 23537395
- [Background] Leasher JL, Bourne RR, Flaxman SR, Jonas JB, Keeffe J, Naidoo K, Pesudovs K, Price H, White RA, Wong TY, Resnikoff S, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global Estimates on the Number of People Blind or Visually Impaired by Diabetic Retinopathy: A Meta-analysis From 1990 to 2010. Diabetes Care. 2016 Sep;39(9):1643-9. doi: 10.2337/dc15-2171. PMID 27555623
- [Background] Klein BE. Overview of epidemiologic studies of diabetic retinopathy. Ophthalmic Epidemiol. 2007 Jul-Aug;14(4):179-83. doi: 10.1080/09286580701396720. PMID 17896294
- [Background] Herman WH, Ali MA, Aubert RE, Engelgau MM, Kenny SJ, Gunter EW, Malarcher AM, Brechner RJ, Wetterhall SF, DeStefano F, et al. Diabetes mellitus in Egypt: risk factors and prevalence. Diabet Med. 1995 Dec;12(12):1126-31. doi: 10.1111/j.1464-5491.1995.tb00432.x. PMID 8750225
- [Background] Alwan A, King H. Diabetes in the eastern Mediterranean region. World Health Stat Q. 1992;45(4):355-9. PMID 1299077
- [Background] Thomas RL, Halim S, Gurudas S, Sivaprasad S, Owens DR. IDF Diabetes Atlas: A review of studies utilising retinal photography on the global prevalence of diabetes related retinopathy between 2015 and 2018. Diabetes Res Clin Pract. 2019 Nov;157:107840. doi: 10.1016/j.diabres.2019.107840. Epub 2019 Nov 14. PMID 31733978
- [Background] Flaxman SR, Bourne RRA, Resnikoff S, Ackland P, Braithwaite T, Cicinelli MV, Das A, Jonas JB, Keeffe J, Kempen JH, Leasher J, Limburg H, Naidoo K, Pesudovs K, Silvester A, Stevens GA, Tahhan N, Wong TY, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global causes of blindness and distance vision impairment 1990-2020: a systematic review and meta-analysis. Lancet Glob Health. 2017 Dec;5(12):e1221-e1234. doi: 10.1016/S2214-109X(17)30393-5. Epub 2017 Oct 11. PMID 29032195
- [Background] Shaikh MZ. Diabetes mellitus--the continuing challenge. J Coll Physicians Surg Pak. 2004 Feb;14(2):63-4. No abstract available. PMID 15228863
- [Background] Tarr JM, Kaul K, Chopra M, Kohner EM, Chibber R. Pathophysiology of diabetic retinopathy. ISRN Ophthalmol. 2013 Jan 15;2013:343560. doi: 10.1155/2013/343560. eCollection 2013. PMID 24563789
- [Background] Wong TY, Mwamburi M, Klein R, Larsen M, Flynn H, Hernandez-Medina M, Ranganathan G, Wirostko B, Pleil A, Mitchell P. Rates of progression in diabetic retinopathy during different time periods: a systematic review and meta-analysis. Diabetes Care. 2009 Dec;32(12):2307-13. doi: 10.2337/dc09-0615. PMID 19940227
- [Background] Sabanayagam C, Yip W, Ting DS, Tan G, Wong TY. Ten Emerging Trends in the Epidemiology of Diabetic Retinopathy. Ophthalmic Epidemiol. 2016 Aug;23(4):209-22. doi: 10.1080/09286586.2016.1193618. Epub 2016 Jun 29. PMID 27355693
- [Background] Elmassry A, Ahmed ISH, Adly N, Torki M. Prevalence of diabetic retinopathy in patients with diabetes in Alexandria and North-West Delta, Egypt. Int Ophthalmol. 2023 Aug;43(8):2883-2895. doi: 10.1007/s10792-023-02692-4. Epub 2023 Mar 24. PMID 36964254